CLINICAL TRIAL: NCT01491230
Title: Neutrophil Extracellular Traps (NETs) Formation Post-hematopoietic Stem Cell Transplantation (HSCT) and Its Relation to Chemotaxis and Creation of Reactive Oxygen Species
Brief Title: Neutrophil Extracellular Traps Formation Post-hematopoietic Stem Cell Transplantation
Acronym: NETs post HSCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Max Planck Institute for Infection Biology (Other); Meir Hospital, Kfar Saba, Israel (Other)
Responsible Party: Principal Investigator, Michal Roll PhD,MBA, Director, Division of Research and Developement, Tel-Aviv Sourasky Medical Center
Other Study IDs: 0443-11-TLV
Record Dates: First submitted 2011-12-11; First posted 2011-12-13 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Childhood Cancer
Keywords: cancer; neutrophil extracellular traps; autologous hematopoietic stem cell transplantation; allogeneic hematopoietic stem cell transplantation; chemotaxis; superoxide production; hydrogen peroxide production; myeloperoxidase
MeSH Terms: conditions — Neoplasms; Chemotaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 10cc of peripheral venous blood will be collected from each patient at several time points: Before transplant, at neutrophil engraftment, 6 weeks, 3 months, 4 months, 6 months, 9 months, 1 year, 1.5 years, 2 years, and 3 years post-transplant, or until normalization of NETs formation in 2 consecutive examinations.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 25 autologous/25 allogeneic patients

SUMMARY:
Identifying the post-transplantation phase wherein neutrophils recover their ability to release NETs could shed new light on the mechanism responsible for the increased susceptibility to infection among these patients and aid in improving their prophylactic antimicrobial treatment. Therefore, we aim to examine neutrophil extracellular traps (NETs) formation, in relation to other neutrophil functions like chemotaxis, superoxide production, hydrogen peroxide production, and the presence of myeloperoxidase, in pediatric patients undergoing autologous and allogeneic hematopoietic stem cell transplantation (HSCT).

DETAILED DESCRIPTION:
Although neutrophil engraftment takes place 10 to 14 days after autologous HSCT, and 15 to 30 days after allogeneic HSCT, using an ablative conditioning regimen, neutrophil dysfunction may persist for longer periods. Relatively scant data exists on neutrophil function following HSCT. After autologous HSCT, the respiratory burst and phagocytosis may be decreased for up to 3 months. After allogeneic HSCT, respiratory burst and chemotaxis are generally decreased for 4 to 6 months. Factors such as continuation of chemotherapy, immunosuppression, and GVHD contribute to this prolonged dysfunction. No data exist on reconstitution of NETs following HSCT.

Nets production and other neutrophil functions will be examined at several time points: before transplantation, at neutrophil engraftment, 6 weeks, 3 months, 6 months, 9 months, 1 year, 1.5 years, 2 years, and 3 years post-transplant, or until normalization of neutrophil function at 2 consecutive time points. Data gathered on patients will cover:

1. Demographics.
2. Tumor histological type, staging, previous chemotherapy regimen, and initial response to treatment.
3. HSCT procedure - type of conditioning regimen, type of graft (autologous or allogeneic - related donor/unrelated donor/cord blood), use of bone marrow stem cells (SCs) or peripheral mobilized SCs, number of SCs given, post-transplant immunosuppression, post-transplant prophylactic antimicrobial treatment, infections during the study period, and GVHD occurrence and treatment.

Neutrophil examinations will be done in collaboration with the Laboratory for Leukocyte Function of the Department of Pediatrics, Meir Medical Center, Kfar Saba and NETs visualization with the Department of Cellular Microbiology at the Max Planck Institute for Infection Biology, Berlin.

ELIGIBILITY:
Inclusion Criteria:

* All infants, children and adolescents undergoing autologous and allogeneic HSCT at the pediatric hemato-oncology departement of Dana children's Hospital.

Exclusion Criteria:

* Severe background diseases (like diabetes and lupus) that there is no data in the literature on their influence on NETs production.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Infants, children and adolescents undergoing autologous and allogeneic HSCT at the pediatric hemato-oncology departement of Dana children's Hospital, Tel-Aviv Sourasky Medical Center, Tel-Aviv, Israel.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sivan Achituv, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Dana Children's Hospital, Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel